CLINICAL TRIAL: NCT05710822
Title: Very High-Power Short-duration Ablation Utilizing the QDOT Micro Ablation Catheter for Pulmonary Vein Isolation - A Multicenter Study.
Brief Title: QDOT Based PVI for Atrial Fibrillation Treatment - The peQasus Study
Acronym: peQasus
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Luebeck (Other)
Responsible Party: Principal Investigator, Christian-H. Heeger, MD, Deputy director, University of Luebeck
Other Study IDs: peQasus study
Record Dates: First submitted 2023-01-17; First posted 2023-02-02 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Atrial Fibrillation
Keywords: Catheter abaltion, very high-power short-duration, QDOT
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: pulmonary vein isolation — pulmonary vein isolation utilizing the QDOT Micro ablation catheter

SUMMARY:
PeQasus is a worldwide, retrospective, multicenter analysis focusing on QDOT based PVI. Data of at least 300 patients with QDOT based PVI will be collected. All data will be evaluated after anonymization. Primary endoints are efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* Suitable for PVI

Exclusion Criteria:

* Non suitable for PVI

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Afib patients with indication to pulmonary vein isolation
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-01-31 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy of the procedure | Periprocedural
  Acute PVI
Saftey (Cardiac tamponade) | Periprocedural
  Periprocedural complications (occurence of cardiac tamponade)
Safety (Stroke) | Periprocedural
  Periprocedural complications (occurence of stroke)
Safety (Bleeding) | Periprocedural
  Periprocedural complications (occurence of puncture site bleeding)

SECONDARY OUTCOMES:
Procedure time | Periprocedural
LA dwelling time | Periprocedural
First pass isolation | Periprocedural
12 months follow-up | 91 days - 12 months after the procedure
  Occurence of aftrial fibrillation or atrial tachycardia >30 Seconds between 91 days and 12 months of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Christian-Hendrik Heeger, MD, Principal Investigator — Department of Rhythmology

IPD SHARING:
Plan to Share IPD: Undecided